CLINICAL TRIAL: NCT05772884
Title: The Potential of Exercise to Reduce Pain and Enhance Mobility in Mid-life Adults Undergoing Opioid Use Treatment
Brief Title: Healthy Aging Through Movement
Acronym: HELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB202002140
Record Dates: First submitted 2023-02-21; First posted 2023-03-16 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use Disorder
Keywords: Pain; Exercise
MeSH Terms: conditions — Opioid-Related Disorders; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: All participants receive the same (single) intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supervised Exercise Intervention (Experimental): Participants will be asked to complete 3 walking sessions per week for 12 weeks. We will ask them to complete at least 1 of these sessions in-person on-site and they will be given the option to complete up to 2 walking sessions per week off-site. Exercise training on-site will be performed on an indoor walking path, 50 min/session (plus 5 min. for each warm-up and cool down).
  Interventions: Other: Supervised Exercise Intervention

INTERVENTIONS:
Other: Supervised Exercise Intervention — Exercise duration will be gradually increased as tolerated to 50 min/session, with intensity ramping up to 65-75% HRmax by week 3. On-site exercise sessions will occur along a pre-marked walking path, and a trained staff member will walk alongside the participant to monitor their heart rate. Speed will be manipulated to achieve desired intensity and to sustain heart rate in the target zone. Heart rate will be monitored and recorded via telemetry during the on-site exercise sessions. Step cadence (i.e., steps/minute) will also be monitored and recorded during the on-site sessions and discussed with participants as a way to understand and track their speed when completing off-site walking sessions on their own.

SUMMARY:
This study aims to examine the effectiveness of a supervised aerobic exercise program for persons with Opioid Use Disorder (OUD). Participants will be enrolled in a 12-week supervised aerobic exercise intervention.

DETAILED DESCRIPTION:
The overall project goals are to test the feasibility and acceptability of our aerobic exercise intervention with this population. Study participation will include a screening and enrollment phase, a baseline assessment, and a 12-week intervention. Participants will be recruited and consented by University of Florida (UF) study staff.

ELIGIBILITY:
Inclusion Criteria:

* Adults must be aged 21-64 years old
* Currently enrolled in OMT (opioid maintenance treatment) or present with at least mild opioid use disorder (endorses at least 2 DSM-V criteria for OUD within a 12-month period),
* Insufficiently physically active (defined as exercising < 20 minutes 3 times/week
* Able to understand and speak English
* Have a body mass index 18.5-40 kg/m^2
* Willing and able to visit research center up to one time time/week for 12 weeks
* Participants will undergo a supervised maximal exercise test and physical exam by medical supervisor to be cleared for participation.

Exclusion Criteria:

* Participants must not have heart disease, or had a stroke, uncontrolled diabetes, thyroid condition an eating disorder
* An uncontrolled major psychiatric condition (e.g., schizophrenia; conditions that are well-controlled, however [e.g., anxiety controlled through therapy] will not be exclusionary), or other medical condition(s) that contraindicate exercise; and may not be participating in a structured exercise training or weight loss program.
* Participants cannot be pregnant; pregnancy is exclusionary
* One individual per household may enroll.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | Baseline up to 4 weeks
  Number of participants screened and enrolled with reasons for ineligibility and non-participation recruitment rate (participants enrolled/month
Intervention adherence | Up to 13 weeks
  Measured as percent study sessions completed on-time (+/- 1 hour of the scheduled session) and the proportion of participants who achieved >75% adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith S Berry, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No